CLINICAL TRIAL: NCT04394533
Title: Does Subarachnoid Administration of Hyperbaric Prilocaine Produce an Improved Recovery From Anaesthesia When Compared With Hyperbaric Bupivacaine When Used to Make Cervical Cerclage Easier in Pregnant Women at Risk of Pre-term Loss?
Brief Title: Hyperbaric Prilocaine Compared With Hyperbaric Bupivacaine in Cervical Cerclage?
Acronym: PRILOCC
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: Obstetric Anaesthetists' Association United Kingdom (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 225703; 2019-001548-23 (EudraCT Number)
Record Dates: First submitted 2020-05-14; First posted 2020-05-19 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Cervical Incompetence in Pregnancy as Antepartum Condition
Keywords: cervical incompetence; cervical cerclage; bupivacaine; prilocaine; subarachnoid block
MeSH Terms: conditions — Uterine Cervical Incompetence | interventions — Prilocaine; Bupivacaine

STUDY DESIGN:
Intervention Model Description: Prospective, parallel group, double-blind, randomised, controlled, superiority trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prilocaine (Intervention) Group (Experimental): Subarachnoid block (SAB) with 40 mg (2 ml) of hyperbaric 20 mg/ml prilocaine and 15 mcg (0.3 ml) fentanyl (50 mcg/ml)
  Interventions: Drug: Prilocaine (Hyperbaric 2%)
- Bupivacaine (Control) Group (Active Comparator): Subarachnoid block (SAB) with 10 mg (2 ml) of hyperbaric 5 mg/ml bupivacaine and 15 mcg (0.3 ml) fentanyl (50 mcg/ml)
  Interventions: Drug: Bupivacaine (Hyperbaric 0.5%)

INTERVENTIONS:
Drug: Prilocaine (Hyperbaric 2%) — 2 ml hyperbaric prilocaine
  Other Names: Hyperbaric prilocaine
  Arms: Prilocaine (Intervention) Group
Drug: Bupivacaine (Hyperbaric 0.5%) — 2 ml hyperbaric bupivacaine
  Other Names: Heavy bupivacaine 0.5%, heavy marcaine 0.5%
  Arms: Bupivacaine (Control) Group

SUMMARY:
Patients that have a "cervical stitch" (cervical cerclage) require an anaesthetic. The most common choice is a spinal block. This is an injection in the back that makes the lower half of the body become temporarily numb and weak. The key aims when choosing which type of anaesthetic are safety for mother and baby, comfort during and after the procedure as well as patient convenience and satisfaction. There are two commonly available choices for the drug used in spinal anaesthesia, bupivacaine and prilocaine. Both have a long history of being safe and effective. One difference observed in studies of these drugs used for spinal anaesthetics in other surgeries is that prilocaine is shorter-acting and it, therefore, takes less time for the return of full strength and sensation of the lower body. This means patients are able to leave hospital sooner and are less likely to need a urinary catheter. The investigators want to see if these benefits can apply to patients having a cervical stitch too, by comparing the recovery of patients having a spinal anaesthetic with one of these two local anaesthetic medications.

DETAILED DESCRIPTION:
Cervical incompetence is defined as the inability to sustain a pregnancy to full term. It is characterized by recurrent second-trimester pregnancy losses. Cervical cerclage is a procedure that is commonly carried out in order to prevent pre-term loss in at-risk pregnancies. The major challenge of performing this as a day case procedure is achieving adequate anaesthesia for comfortable performance of the cerclage whilst providing adequate regression of motor and sensory blocks to allow ambulation and bladder control within an appropriate timescale. Spinal anaesthesia, or subarachnoid block (SAB), is commonly employed to facilitate a wide variety of pelvic and lower limb surgeries. In the United Kingdom, the commonly administered subarachnoid agents are bupivacaine, prilocaine and, until recent decades, lidocaine. The duration of action of bupivacaine makes it less well suited to day surgery as it is often difficult to reach discharge criteria within a convenient time frame. The investigators aim to examine the recovery profiles of two equipotent doses of hyperbaric prilocaine and bupivacaine. Given the evidence, the survey of practice in other centres and the commonly used doses at this institution the following regimens will be compared:

* 40 mg of hyperbaric 2% prilocaine with 15 mcg of fentanyl (intervention) and
* 10 mg of hyperbaric 0.5% bupivacaine with 15 mcg of fentanyl (comparator).

Primary Objective:

This study aims to determine if a difference exists between the time required for regression of motor block between two commonly used and equipotent doses of subarachnoid hyperbaric prilocaine and bupivacaine.

* The hypothesis is that SAB with hyperbaric 2% prilocaine will result in a clinically significant reduction in time taken for regression of motor blockade, as determined by achieving a Bromage score* of I, when compared to an equipotent dose of hyperbaric bupivacaine when used to facilitate cervical cerclage in pregnant women in the second trimester of pregnancy.
* The null hypothesis is that no clinically significant difference exists while the alternative hypothesis is that such a difference truly exists.

Secondary Objectives:

* To compare the intraoperative characteristics of the subarachnoid block and quality of intraoperative anaesthesia in the two groups.
* To compare the recovery profiles in the two groups
* To compare the incidence of complications in the two groups
* To compare the satisfaction of the participants in each group This is a prospective, single centre, parallel group, double-blind, randomised, controlled, superiority trial. The sample size will consist of 135 patients having elective cervical cerclage, under SAB, due to cervical incompetence.

Sample Size Calculation The primary outcome measurement is the comparison of the difference in time taken for regression of lower limb motor block with hyperbaric (heavy) 2% prilocaine compared to hyperbaric (heavy) 0.5% bupivacaine. Assuming, based on pilot data, that the time to regression of motor block has a standard deviation of up to 60 mins; complete data on 128 participants (64 to each arm) would give 80% power to detect a plausible and clinically important 30-min difference between groups at the 0.05 significance level. To allow for up to 5% dropout, the study will recruit 135 women.

Random allocation to groups will be achieved using "Castor" randomisation software. The sequence will have been previously determined, prior to recruitment, using computer software, by random permuted blocks. Subsequently, the subjects who give written informed consent will be randomly assigned a unique 3-digit subject number. The subject number together uniquely identifies every subject eligible for the study. Randomisation will take place on the day of surgery by a non-operating healthcare professional who will randomise according to the "Castor" software. If code breaking is necessary, this will be done by pharmacy. As soon as 128 evaluable subjects have been included in the study, recruitment will be stopped.

Analysis After checking for normality by standard diagnostic plots, a comparison between the groups will be made using multiple regression with a dummy variable for treatment arm. A correction will be made for unequal variance using the robust standard errors. Adjustment will be made for maternal BMI and height, as these are known to be related to anaesthetic effect.

No power calculation has been carried out for the secondary outcomes, and no priority is made between them. Continuous measures, including the patient satisfaction score, will be analysed as described above for the primary outcome. Binary measures will be expressed as percentages, and compared by means of risk ratios, using binary regression with a log link, adjusted for BMI and height, as described above.

Subgroup analyses: A comparison will be made between normal weight and obese women (BMI over 30 kg.m-2); and between women above and below 165 cm in height, using an interaction test to check for a difference in treatment effect.

No interim analysis is planned.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (ASA score 2 or 3) pregnant women presenting for elective cervical cerclage under SAB.
* Age > 18 years

Exclusion Criteria:

* Inability to read or understand the patient information sheet (PIS)
* Age < 18 years
* Unable or unwilling to consent to participation
* non-elective procedure
* serious co-morbidities (ASA score 4 or above)
* any contraindication to SAB, e.g. local or generalised infection, active central nervous system disease, coagulation disorders or anti-coagulant medication
* any history of allergic reaction to any of the medications in the protocol
* concomitant use of class III anti-arrhythmics (sulfonamides, antimalarials, sodium nitroprussate, nitroglycerin, other local anaesthetics)
* any contraindication to the use of bupivacaine or prilocaine as listed in the SmPCs.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2021-08-27 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Time from SAB to Bromage score of I | 24 hours
  Difference in time taken for regression of lower limb block between the two groups

SECONDARY OUTCOMES:
Time from SAB until loss of cold sensation to ethyl chloride spray at tenth thoracic dermatomal level (T10) | 30 minutes
  Difference in time (minutes) for loss of cold sensation at tenth thoracic dermatomal level (T10)
Time from SAB until motor block Bromage IV | 30 minutes
  Difference in time take for complete motor block to occur
Determine uppermost level of sensory block | 20 minutes
  Determine uppermost (cephalad) dermatomal level of sensory block as measured by loss of cold sensation to ethyl chloride spray at 20 minutes (mean).
Degree of motor block | 20 minutes
  Mean degree of motor block as assessed on the Bromage scale at 20 minutes (from I-IV)
Maximum intraoperative Numerical Rating Score (NRS) [0-10] | 1 hour
  Mean pain score on the NRS (from 0-10) of maximal discomfort experienced during the procedure
Time from SAB to ambulation | 24 hours
  Mean time in minutes from SAB to ambulation
Time from SAB to micturition | 24 hours
  Mean time in minutes from SAB to micturition
Time from SAB to discharge | 24 hours
  Mean time in minutes from SAB to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Desire Onwochei, MBBS, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No